CLINICAL TRIAL: NCT07100535
Title: Education and Literacy for an Active Life
Brief Title: Education and Literacy for an Active Life (Educação e Literacia Para Uma Vida Ativa)
Acronym: ELeVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lusofona University (Other)
Collaborators: Faculty of Medicine of Universidade de Lisboa (FMUL) (Unknown)
Responsible Party: Principal Investigator, António Videira-Silva, Professor, Lusofona University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FEFD16012024
Record Dates: First submitted 2025-07-16; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Health Literacy; Physical Activity; Nutrition; Sedentary Behaviors; Sleep; Mental Health
Keywords: Health literacy; Nutrition; Physical activity; Sedentary behaviours; Sleep; Mental health
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Psychological Well-Being | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Phase 1. Open label. Intervention and assessments will be performed by the core researchers.
  Phase 2. Intervention will be applied by trained professors (not part of the research team). Assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and Literacy for an Active Life (Experimental): Participants will be exposed to 50-minute sessions (only four sessions in Phase 1), targeting health literacy (across the four dimensions: access, comprehension, evaluation and application) on nutrition, sedentary behaviour, physical activity, sleep and mental health. Sessions will use interactive and student-centred methodologies, such as discussions, videos, practical activities, and group work, to promote participation and active learning. The intervention will be implemented uniformly across schools with the support of teachers. Activities will be adapted to the school context and age group to ensure feasibility and relevance.
  Interventions: Behavioral: Education and Literacy for an Active Life
- Standard School Curriculum (No Intervention): Participants will not receive the health literacy intervention during the study period, receiving only standard school curriculum.

INTERVENTIONS:
Behavioral: Education and Literacy for an Active Life — This study will assess the effectiveness of a school-based health literacy intervention on the four dimensions of health literacy (i.e., access, understanding, evaluation, and application) on diet, sedentary behaviour, physical activity, sleep, and mental health in 5th and 6th graders (aged 9-12), and explored its implementation feasibility.
  Other Names: Educação e Literacia para uma Vida Ativa
  Arms: Education and Literacy for an Active Life

SUMMARY:
Health literacy is essential for children to develop healthy behaviors that persist into adulthood. It enables the access, understanding, evaluation, and application of health-related information, being a key component of health education.

This study was designed as a randomized controlled study, aiming to analyze the effectiveness and feasibility of a school intervention to improve health literacy of 5th and 6th grade students on nutrition, physical activity, sleep, and mental health. Intervention will be delivered in two phases. Phase 1 will involve a pilot intervention comprising four sessions conducted over a three-month period in two schools representing distinct socioeconomic contexts. Phase 2 will scale the intervention nationally, expanding to include additional schools across Portugal. This phase will include eight sessions conducted over one entire school-year (September-June), and will integrate adjustments based on the limitations and insights identified during the pilot study. Phase 2 will additionally include 20-month follow-up assessments to be performed at the end of the following school-year (20-month).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the classes of the included schools
* Agreed to participate
* Informed consent/assent signature

Exclusion Criteria:

* Severe cognitive or learning disabilities (significant impairment of the ability to engage with the intervention content or complete assessment tools)
* Absenteeism (missing ≥30% of the scheduled sessions)
* Concurrent participation in similar interventions (concurrent enrolment in other structured health, nutrition, or mental health programs that could confound study results)

Note: students with medical conditions that limit their ability to participate in physical activities will not be excluded. The presence of such conditions will be further considered in the analysis.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Overall health literacy score | Data will be assessed at baseline (before randomisation), at the end of the intervention (for Phase 1: 3-month; for Phase 2: end of the academic year, 8-month) and at follow-up (Phase 2-only: at the end of the following academic year, 20-month).
  Overall health literacy score, assessed by the Questionnaire on Literacy in Health Behaviours for Children (QLCS-C), specifically developed for this study and adapted to the Portuguese educational and sociocultural context. This instrument is under validation and was designed to evaluate health literacy competences in children aged 9-12 years, encompassing four core health literacy dimensions: access, comprehension, evaluation and application, of health-related information. The instrument covers five critical domains of health promotion relevant to this age group: diet, PA, sedentary behaviour, sleep and mental health and includes a total of 47 items, scored 0-20 points/item, on a total of 0-100 points). The higher the score, the higher the Literacy level. Item development was based on an extensive review of validated instruments and international guidelines.

SECONDARY OUTCOMES:
Health Literacy on Nutrition | Data will be assessed at baseline (before randomisation), at the end of the intervention (for Phase 1: 3-month; for Phase 2: end of the academic year, 8-month) and at follow-up (Phase 2-only: at the end of the following academic year, 20-month).
  Health Literacy on Nutrition will be assessed by the Questionnaire on Literacy in Health Behaviours for Children (QLCS-C). Items on Nutrition (1-20/47) reflect core principles of food literacy and public health nutrition, including nutrient awareness, label reading, and balanced eating habits. Along with categorical analysis, numerical analysis will be also performed (score 0-20). The higher the score, the higher the Literacy level.
Health Literacy on Physical Activity | Data will be assessed at baseline (before randomisation), at the end of the intervention (for Phase 1: 3-month; for Phase 2: end of the academic year, 8-month) and at follow-up (Phase 2-only: at the end of the following academic year, 20-month).
  Health Literacy on Physical Activity will be assessed by the Questionnaire on Literacy in Health Behaviours for Children (QLCS-C). Items on Physical Activity (21-30/47) include an adaptation from the Physical Activity Questionnaire for Adolescents - PAQ-A (Kowalski et al., 2004) focusing on knowledge, perceived benefits, obstacles, and engagement in activity. Along with categorical analysis, numerical analysis will be also performed (score 0-20). The higher the score, the higher the Literacy level.
Health Literacy on Sedentary Behaviour | Data will be assessed at baseline (before randomisation), at the end of the intervention (for Phase 1: 3-month; for Phase 2: end of the academic year, 8-month) and at follow-up (Phase 2-only: at the end of the following academic year, 20-month).
  Health Literacy on Sedentary Behaviour will be assessed by the Questionnaire on Literacy in Health Behaviours for Children (QLCS-C). Items on Sedentary Behaviour (31-33/47) draws from the Adolescent Sedentary Activity Questionnaire - ASAQ (Hardy et al., 2007), adapted to assess screen time and perceived health impacts. Along with categorical analysis, numerical analysis will be also performed (score 0-20). The higher the score, the higher the Literacy level.
Health Literacy on Sleep | Data will be assessed at baseline (before randomisation), at the end of the intervention (for Phase 1: 3-month; for Phase 2: end of the academic year, 8-month) and at follow-up (Phase 2-only: at the end of the following academic year, 20-month).
  Health Literacy on Sleep will be assessed by the Questionnaire on Literacy in Health Behaviours for Children (QLCS-C). Items on Sleep (34-41/47) were specifically developed for this study, informed by international public health guidelines on sleep hygiene in childhood (Paruthi et al., 2016). These items explore the children's understanding of sleep routines, behaviours, caffeine use, and reliable sources of information on sleep. Although thematically related to constructs evaluated in clinical tools such as the Pittsburgh Sleep Quality Index (Pittsburgh Sleep Quality Index - PSQI (Buysse et al., 1989), the purpose of these items is educational, aligned with health literacy competences, and adapted to children's cognitive levels. Along with categorical analysis, numerical analysis will be also performed (score 0-20). The higher the score, the higher the Literacy level.
Health Literacy on Mental Health | Data will be assessed at baseline (before randomisation), at the end of the intervention (for Phase 1: 3-month; for Phase 2: end of the academic year, 8-month) and at follow-up (Phase 2-only: at the end of the following academic year, 20-month).
  Health Literacy on Mental health will be assessed by the Questionnaire on Literacy in Health Behaviours for Children (QLCS-C). Items on Mental Health (42-47/47) focus on emotional literacy, stress regulation, and social support, with two items adapted from the Flourishing Scale (Diener et al., 2009). Along with categorical analysis, numerical analysis will be also performed (score 0-20). The higher the score, the higher the Literacy level.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Lusófona - Centro Universitário Lisboa, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Paruthi S, Brooks LJ, D'Ambrosio C, Hall WA, Kotagal S, Lloyd RM, Malow BA, Maski K, Nichols C, Quan SF, Rosen CL, Troester MM, Wise MS. Recommended Amount of Sleep for Pediatric Populations: A Consensus Statement of the American Academy of Sleep Medicine. J Clin Sleep Med. 2016 Jun 15;12(6):785-6. doi: 10.5664/jcsm.5866. PMID 27250809
- [Background] Sirajudeen MS, Waly M, Manzar MD, Alqahtani M, Alzhrani M, Alanazi A, Unnikrishnan R, Muthusamy H, Saibannavar R, Alrubaia W. Physical activity questionnaire for older children (PAQ-C): Arabic translation, cross-cultural adaptation, and psychometric validation in school-aged children in Saudi Arabia. PeerJ. 2022 Apr 12;10:e13237. doi: 10.7717/peerj.13237. eCollection 2022. PMID 35433134
- [Background] Hardy LL, Booth ML, Okely AD. The reliability of the Adolescent Sedentary Activity Questionnaire (ASAQ). Prev Med. 2007 Jul;45(1):71-4. doi: 10.1016/j.ypmed.2007.03.014. Epub 2007 Apr 14. PMID 17532371